CLINICAL TRIAL: NCT05862935
Title: Influence of Physical Exercise as Adjuvant Treatment in Patients With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Asociación de Familiares de Alzheimer de Valladolid (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI-DOC002-ALP
Record Dates: First submitted 2023-05-03; First posted 2023-05-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Physical exercise; Locomotion
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The persons analyzing the data collected (investigators, statician) will not know to which group each person belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Physical Activity (Phase I: Strength training; Phase II: AMRAP training) (Experimental): These patients, in addition to receiving the usual treatment for their pathology, carry out supervised activity consisting of:
  * Warm-up
  * Strength circuit; At phase I it will be a standard strength training, while at Phase 2 it will be an AMRAP training)
  Interventions: Other: Supervised Physical Activity (AMRAP -As Many Repetitions As Possible): Phase 2; Other: Supervised Physical Activity: Phase 1
- Control (No Intervention): These patients only receive the usual treatment for their pathology.

INTERVENTIONS:
Other: Supervised Physical Activity (AMRAP -As Many Repetitions As Possible): Phase 2 — 20-30 min/session, 3 times/week for 4 weeks. After a 5-min warm-up, participants perform a moderate-intensity functional training program. This program is designed in circuit mode consisting of 6 global functional exercises: i) sit and stand, ii) forward lunges, iii) chest press, iv) high row, v) lateral shoulder raises and vi) heel raises. Participants must complete the highest number of repetitions and/or rounds as possible (AMRAP) in 15-min without a designated rest.
  Other Names: AMRAP intervention
  Arms: Supervised Physical Activity (Phase I: Strength training; Phase II: AMRAP training)
Other: Supervised Physical Activity: Phase 1 — 40-60 min/session, 3 times/week for 12 weeks. After a 5-min warm-up, participants performed 6 global functional exercises: i) sit-to-stand; ii) chest press, iii) forward lunges; iv) unilateral shoulder raises; v) unilateral row; and vi) heel raises. The initial volume is 2 sets and 8 repetitions and it will progressively increase until 3 sets and 12 repetitions.
  Other Names: Basic strength intervention
  Arms: Supervised Physical Activity (Phase I: Strength training; Phase II: AMRAP training)

SUMMARY:
The goal of this non-randomized clinical trial is to assess the effects of strength training in the physical function of Alzheimer's disease (AD) patients. The main question it aims to answer are:

1. Is a basic strength training enough to improve physical function in AD patients?
2. Is an exercise intervention able to delayed the progression of the disease?
3. Is an AMRAP intervention feasible in AD patients?

Participants in the exercise group will perform a 16-weeks program divided in two phases (phase 1: basic strength training; phase 2: AMRAP training). Participants in both (exercise and control) groups will receive their usual care treatments which include occupational therapy, musicotherapy, cognitive stimulation and sensory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* MMSE (Mini-Metal State Examination) score of ≥15 out of 35 (at screening less than 2 months prior to baseline visit)
* Age ≥60 years old
* Be able to walk with or without aids
* Be able to follow verbal instructions

Exclusion Criteria:

* Surgery in the last 3 months
* Exhibit clear signs of disorientation
* Clinically confirmed signs of aggressiveness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | 0 weeks, 12 weeks, 16 weeks of intervention. 8 weeks of detraining
  Changes in the SPPB Score (Short Physical Performance Battery; Range between 0 "worst performance" and 12 "best performance")

SECONDARY OUTCOMES:
Handgrip strength | 0 weeks, 12 weeks, 16 weeks of intervention. 8 weeks of detraining
  Changes in the hang-up strength in the dominant side
Body mass index | 0 weeks, 12 weeks, 16 weeks of intervention. 8 weeks of detraining
  Changes in the body mass index
Practicability of AMRAP (As Many Repetitions As Possible) training; it will be analysed by calculating both intra- and inter-subject coefficient variation. | Every session (during 13 sessions)
  This variable evaluates the applicability of this tipe of training in patients with Alzheimer disease

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea Miguel de Cervantes, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No